CLINICAL TRIAL: NCT04301986
Title: Patient Acceptance and Preference Among Screening Modalities for Detection of Barrett's Esophagus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: American Gastroenterological Association (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-3290
Record Dates: First submitted 2020-02-24; First posted 2020-03-10 (Actual); Results first posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2022-09

CONDITIONS: Barrett Esophagus; GERD
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux | interventions — Endoscopes; Endoscopy, Digestive System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TNE Followed by EGD (Experimental): Subjects will undergo administration of a transnasal endoscopy (TNE) prior to their scheduled clinically indicated upper endoscopy performed per routine standard of care. Following the procedure, a follow-up phone call will be made during which an impact of events scale related to the subjective distress of each procedure, a preference and acceptance questionnaire, and adverse events related to study participation will be collected.
  Interventions: Device: Transnasal Endoscopy (TNE); Device: Esophagogastroduodenoscopy
- Cytosponge, then TNE, followed by EGD (Experimental): Subjects will undergo administration of Cytosponge and transnasal endoscopy (TNE) prior to their scheduled clinically indicated upper endoscopy performed per routine standard of care. Following the procedure, a follow-up phone call will be made during which an impact of events scale related to the subjective distress of each procedure, a preference and acceptance questionnaire, and adverse events related to study participation will be collected.
  Interventions: Device: Cytosponge; Device: Transnasal Endoscopy (TNE); Device: Esophagogastroduodenoscopy

INTERVENTIONS:
Device: Cytosponge — In a seated position, subjects will swallow the Cytosponge capsule with 150-250 mL of water. Seven minutes and 30 seconds to ten minutes after ingestion, the sponge is then withdrawn by gentle traction on the suture. After retrieval, the string is cut and the retrieved foam sphere containing the cytological specimen is immersed in fixative and stored refrigerated (1° to 12°C [34° to 54°F]).
  Other Names: Cytosponge Cell Collection Device
  Arms: Cytosponge, then TNE, followed by EGD
Device: Transnasal Endoscopy (TNE) — In an upright position, the scope will be inserted via the nares to examine the posterior pharynx, esophagus and proximal stomach with the transnasal endoscopy approach. The scope will be withdrawn from the nares following completion of the exam.
  Other Names: Olympus Neonatal (ultrathin) endoscope
Device: Esophagogastroduodenoscopy — Laying on the subjects' left side, the flexible endoscope is inserted through the mouth to allow visualization of the esophageal mucosa from the upper esophageal sphincter all the way to the esophagogastric junction (EGJ).
  Other Names: EGD

SUMMARY:
To assess patient acceptance and preference among screening modalities, Esophagogastroduodenoscopy (EGD), Transnasal Esophagoscopy (TNE), and Cytosponge for Barrett's esophagus (BE). Subjects will undergo administration of Cytosponge and transnasal endoscopy (TNE) prior to their scheduled clinically indicated upper endoscopy performed per routine standard of care. Following the procedure, a follow-up phone call will be made during which an impact of events scale related to the subjective distress of each procedure, a preference and acceptance questionnaire, and adverse events related to study participation will be collected.

DETAILED DESCRIPTION:
Potential subjects will be identified via protocol and Institutional Review Board (IRB) methods prior to obtaining written informed consent. Once written informed consent is obtained and baseline demographic and medical history is collected, subjects will undergo administration of Cytosponge and transnasal endoscopy (TNE) prior to their scheduled clinically indicated upper endoscopy performed per routine standard of care. Following the procedure, a follow-up phone call will be made during which an impact of events scale related to the subjective distress of each procedure, a preference and acceptance questionnaire, and adverse events related to study participation will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one of the following: Gastroesophageal Reflux Disease (GERD) OR Barrett's esophagus (BE)
* At least 18 years of age at time of consent
* Able and willing to provide written informed consent
* Able and willing to comply with required study procedures and follow-up schedule
* Presenting to UNC Hospitals for routine care upper endoscopy

Exclusion Criteria:

* History of pre-existing esophageal stenosis/ stricture, esophageal diverticulum or significant esophageal anatomic abnormalities (masses, obstructive lesions, etc.)
* History of head and neck malignancy or anatomical abnormalities of the nasopharynx
* Any history of Ear, Nose and Throat (ENT) surgery
* History of significant epistaxis or hereditary hemorrhagic telangiectasia (HHT)
* Sinus or pulmonary infection in the last 4 weeks
* Current use of blood thinners such as coumadin, warfarin, clopidogrel, heparin and/or low molecular weight heparin (requires discontinuation of medication 7 days prior to and 7 days after esophagogastroduodenoscopy [EGD] and Cytosponge administration, aspirin use is OK).
* Known bleeding disorder
* Pregnancy, or planned pregnancy during the course of the study.
* Any history of esophageal varices, liver impairment of moderate or worse severity (Child's- Pugh class B & C) or evidence of varices noted on any past endoscopy
* Any history of esophageal surgery, except for uncomplicated fundoplication
* History of coagulopathy, with international normalised ratio (INR) >1.3 and/or platelet count of <75,000
* General poor health, multiple co-morbidities placing the patient at risk, or otherwise unsuitable for trial participation
* Subject has any condition that, in the opinion of the investigator or sponsor, would interfere with accurate interpretation of the study objectives or preclude participation in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Swathi Eluri, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- TNE Followed by EGD: Participants will undergo administration of a transnasal endoscopy (TNE) prior to their scheduled clinically indicated upper endoscopy performed per routine standard of care. Following the procedure, a follow-up phone call will be made during which an impact of events scale related to the subjective distress of each procedure, a preference and acceptance questionnaire, and adverse events related to study participation will be collected.
  Transnasal Endoscopy (TNE): In an upright position, the scope will be inserted via the nares to examine the posterior pharynx, esophagus and proximal stomach with the transnasal endoscopy approach. The scope will be withdrawn from the nares following completion of the exam.
  Esophagogastroduodenoscopy: Laying on the participants' left side, the flexible endoscope is inserted through the mouth to allow visualization of the esophageal mucosa from the upper esophageal sphincter all the way to the esophagogastric junction (EGJ).
- Cytosponge, Then TNE, Followed by EGD: Participants will undergo administration of Cytosponge and transnasal endoscopy (TNE) prior to their scheduled clinically indicated upper endoscopy performed per routine standard of care. Following the procedure, a follow-up phone call will be made during which an impact of events scale related to the subjective distress of each procedure, a preference and acceptance questionnaire, and adverse events related to study participation will be collected.
  Cytosponge: In a seated position, participants will swallow the Cytosponge capsule with 150-250 mL of water. Seven minutes and 30 seconds to ten minutes after ingestion, the sponge is then withdrawn by gentle traction on the suture. After retrieval, the string is cut and the retrieved foam sphere containing the cytological specimen is immersed in fixative and stored refrigerated (1° to 12°C [34° to 54°F]).
  Transnasal Endoscopy (TNE): In an upright position, the scope will be inserted via the nares to examine the posterior pharynx, esophagus and proximal stomach with the transnasal endoscopy approach. The scope will be withdrawn from the nares following completion of the exam.
  Esophagogastroduodenoscopy: Laying on the participants' left side, the flexible endoscope is inserted through the mouth to allow visualization of the esophageal mucosa from the upper esophageal sphincter all the way to the esophagogastric junction (EGJ).
Period: Overall Study
Arm/Group | TNE Followed by EGD | Cytosponge, Then TNE, Followed by EGD
Started | 0 | 24
Completed | 0 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants enrolled into the arm completing all 3 maneuvers (i.e., Cytosponge, Then TNE, Followed by EGD).
Groups:
- Total: Total of all reporting groups
Arm/Group | TNE Followed by EGD | Cytosponge, Then TNE, Followed by EGD | Total
Number analyzed (Participants) | 0 | 24 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 12 | 12
  >=65 years |  | 12 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 5 | 5
  Male |  | 19 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 24 | 24
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States |  | 24 | 24

OUTCOME MEASURES:

1. Primary Outcome: 7 Days Post-EGD Impact of Events Score (IES)
Description: Impact of Events Score (IES): scale was developed to assess the distress associated with a specific life event. IES scores range from 0-75, with higher scores indicating more severe distress associated from an event. Scores ≥ 44 indicate a event has severe impact on self-reported distress while scores ≤ 25 indicate the event may have an effect on distress.
Time Frame: 7 days post-EGD
Population: All participants enrolled into the arm completing all 3 maneuvers (i.e., Cytosponge, Then TNE, Followed by EGD).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cytosponge: Participants will undergo administration of Cytosponge.
  Cytosponge: In a seated position, participants will swallow the Cytosponge capsule with 150-250 mL of water. Seven minutes and 30 seconds to ten minutes after ingestion, the sponge is then withdrawn by gentle traction on the suture. After retrieval, the string is cut and the retrieved foam sphere containing the cytological specimen is immersed in fixative and stored refrigerated (1° to 12°C [34° to 54°F]).
- Transnasal Endoscopy (TNE): Participants will undergo administration of TNE. Transnasal Endoscopy (TNE): In an upright position, the scope will be inserted via the nares to examine the posterior pharynx, esophagus and proximal stomach with the transnasal endoscopy approach. The scope will be withdrawn from the nares following completion of the exam.
- Esophagogastroduodenoscopy (EGD): Esophagogastroduodenoscopy: Laying on the participants' left side, the flexible endoscope is inserted through the mouth to allow visualization of the esophageal mucosa from the upper esophageal sphincter all the way to the esophagogastric junction (EGJ).
Arm/Group | TNE Followed by EGD | Cytosponge | Transnasal Endoscopy (TNE) | Esophagogastroduodenoscopy (EGD)
Number analyzed (Participants) | 0 | 24 | 24 | 24
units on a scale |  | 1.42 (2.89) | 1.21 (2.54) | 0 (0)

2. Secondary Outcome: Visual Analog Scale (VAS) Score
Description: Visual Analog Scale (VAS): 100-mm horizontal line on which the participant's pain intensity is represented by a point between the extremes of 0 reflecting "no pain at all" and 100 reflecting the "worst pain imaginable."
Time Frame: Day 1, Post-procedure (<24 hours of procedure completion)
Population: All participants enrolled into the arm completing all 3 maneuvers (i.e., Cytosponge, Then TNE, Followed by EGD).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TNE Followed by EGD | Cytosponge | Transnasal Endoscopy (TNE) | Esophagogastroduodenoscopy (EGD)
Number analyzed (Participants) | 0 | 23 | 23 | 24
units on a scale |  | 14.69 (15.69) | 49.57 (28.72) | 5.5 (11.59)

3. Secondary Outcome: 7 Days Post-EGD Willingness to Repeat
Description: 7 days post-EGD participants were asked about their willingness to repeat the maneuvers (Yes/No).
Time Frame: 7 days post-EGD
Population: All participants enrolled into the arm completing all 3 maneuvers (i.e., Cytosponge, Then TNE, Followed by EGD).
Measure: Count of Participants; unit: Participants
Arm/Group | TNE Followed by EGD | Cytosponge | Transnasal Endoscopy (TNE) | Esophagogastroduodenoscopy (EGD)
Number analyzed (Participants) | 0 | 24 | 24 | 24
Participants
  Yes |  | 24 | 21 | 24
  No |  | 0 | 3 | 0

4. Secondary Outcome: 7 Days Post-EGD Ranking of Preferred Screening Modality
Description: Participants asked to rank preferred screening modality in order (1,2,3). Scores range from 0-3. Scores of 1 indicate a preference, while scores of 3 indicate aversion.
Time Frame: 7 days post-EGD
Population: Preferred screening was inadvertently omitted during form creation and these data were not collected.
Arm/Group | TNE Followed by EGD | Cytosponge | Transnasal Endoscopy (TNE) | Esophagogastroduodenoscopy (EGD)
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants Reporting Preferred Screening Modality
Description: Participants asked "Which procedure would you prefer to undergo again?" Only one item could be selected.
Time Frame: 7 days post-EGD
Population: All participants enrolled into the arm completing all 3 maneuvers (i.e., Cytosponge, Then TNE, Followed by EGD).
Measure: Count of Participants; unit: Participants
Groups:
- Cytosponge, Then TNE, Followed by EGD: Participants will undergo administration of Cytosponge and transnasal endoscopy (TNE) prior to their scheduled clinically indicated upper endoscopy performed per routine standard of care. Following the procedure, a follow-up phone call will be made during which an impact of events scale related to the subjective distress of each procedure, a preference and acceptance questionnaire, and adverse events related to study participation will be collected.
  Cytosponge: In a seated position, subjects will swallow the Cytosponge capsule with 150-250 mL of water. Seven minutes and 30 seconds to ten minutes after ingestion, the sponge is then withdrawn by gentle traction on the suture. After retrieval, the string is cut and the retrieved foam sphere containing the cytological specimen is immersed in fixative and stored refrigerated (1° to 12°C [34° to 54°F]).
  Transnasal Endoscopy (TNE): In an upright position, the scope will be inserted via the nares to examine the posterior pharynx, esophagus and proximal stomach with the transnasal endoscopy approach. The scope will be withdrawn from the nares following completion of the exam.
  Esophagogastroduodenoscopy: Laying on the subjects' left side, the flexible endoscope is inserted through the mouth to allow visualization of the esophageal mucosa from the upper esophageal sphincter all the way to the esophagogastric junction (EGJ).
Arm/Group | TNE Followed by EGD | Cytosponge, Then TNE, Followed by EGD
Number analyzed (Participants) | 0 | 24
Participants
  Cytosponge |  | 6
  TNE |  | 1
  EGD |  | 17

6. Secondary Outcome: Factors Influencing the Preferred Screening Modality
Description: Participants asked what factors influenced preference in choosing preferred screening modality. Selection options were: discomfort/pain; time (preparation time and post-procedure); cost; and sedation. Participants could provide multiple response selections.
Time Frame: 7 days post-EGD
Population: All participants enrolled into the arm completing all 3 maneuvers (i.e., Cytosponge, Then TNE, Followed by EGD).
Measure: Count of Participants; unit: Participants
Arm/Group | TNE Followed by EGD | Cytosponge, Then TNE, Followed by EGD
Number analyzed (Participants) | 0 | 24
Participants
  Discomfort/pain |  | 12
  Time |  | 6
  Cost |  | 3
  Sedation |  | 13
  Other |  | 4

ADVERSE EVENTS:
Time Frame: From the time of informed consent through seven days post-intervention, a total of 8 days.
Description: All procedures were completed sequentially during the same visit with study staff inquiring about the occurence of adverse events following completion of all procedures. Thus, determination of which particular device to which an event might be attributable is not possible.
Arm/Group | TNE Followed by EGD | Cytosponge, Then TNE, Followed by EGD
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/24
Other Adverse Events (participants affected / at risk) | 0/0 | 3/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TNE Followed by EGD (N=0) | Cytosponge, Then TNE, Followed by EGD (N=24)
Pain - Throat/Esophageal (Gastrointestinal disorders) | 0 | 3 (3) — Pain experienced in the throat/esophagus

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT04301986/Prot_SAP_001.pdf